CLINICAL TRIAL: NCT02539914
Title: Interactive System for Diagnostics and Rehabilitation of Cognitive-motor Deficits: Controlled Longitudinal Clinical Study With Stroke Patients
Brief Title: Feasibility Study of a Virtual Reality Cognitive-motor Task Based on Positive Stimuli for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Serviço de Saúde da Região Autónoma da Madeira (SESARAM), E.P.E. (Unknown)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Professor Auxiliar, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 303891- 47/2013
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: Virtual reality; Motor and cognitive rehabilitation; Positive emotion stimuli
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VR motor-cognitive task (Experimental): The VR motor-cognitive task group will perform a virtual reality motor and cognitive attention/memory task customized to each user in terms of the positive content.
  Interventions: Other: Virtual Reality
- Standard rehabilitation (Active Comparator): The standard rehabilitation group will perform conventional motor and cognitive rehabilitation tasks.
  Interventions: Other: Standard

INTERVENTIONS:
Other: Virtual Reality — Virtual reality based upper-limb motor and cognitive task
  Arms: VR motor-cognitive task
Other: Standard — Standard upper-limb motor and cognitive rehabilitation tasks
  Arms: Standard rehabilitation

SUMMARY:
The purpose of this study is to determine whether it is feasible to use a virtual reality task for stroke rehabilitation for training motor and cognitive (attention and memory) domains based on the use of positive stimuli, and to evaluate the potential benefits in comparison to standard rehabilitation.

DETAILED DESCRIPTION:
There is evidence that positive emotion stimuli can lead to improved performance in attention tasks and the investigators aim to understand the benefits of using this principle in cognitive and upper-limb motor rehabilitation following stroke. For this purpose, the investigators developed a VR attention task in which the user has to find a target image within a variable number of distractors by controlling a virtual arm. In some levels of the task the target has to be memorized, hence training both attention and memory. The target stimuli are positive images based on the individual preferences of each user.

40 participants within the first 6 months after stroke will be randomly allocated to one of two groups: 1) VR motor-cognitive task or 2) standard rehabilitation. The VR motor-cognitive task group will use the above described virtual task customized to each user in terms of the positive content. This also includes selected music that will be introduced in half of the sessions. The standard rehabilitation group will undergo conventional motor and cognitive rehabilitation. The intervention consists of 12 sessions of 45 minutes administered within a 4-6 weeks period. The participants will be evaluated using a number motor and cognitive assessment scales at baseline, end of the intervention and a 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke within the first 6 months post-stroke
* motor impairment of the upper extremity but with a minimum score of 28 in the Motricity Index (elbow flexion and shoulder abduction domains combined score)
* cognitive deficit but with enough capacity to understand the task and follow instructions with a minimum score of 11 over 17 in the Token Test (6-item version, portuguese population)
* able to read

Exclusion Criteria:

* previous motor and/or cognitive deficits
* normal cognitive functioning with a score above 26 points in the Montreal Cognitive Assessment
* unilateral spatial neglect
* moderate to severe depressive symptomatology with a score above 20 points in the Geriatric Depression Scale
* vision disorders that may interfere with the execution of the task

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Fugl-Meyer Assessment Test (upper extremity) | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in motor and joint functioning of the paretic upper extremity.
Change form baseline in the Chedoke Arm and Hand Activity Inventory | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in the functionality of the paretic upper extremity.
Change from baseline in the Montreal Cognitive Assessment | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.

SECONDARY OUTCOMES:
Change from baseline in the Barthel Index | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in independence in activities of daily living.
Change from baseline in the Modified Ashworth Scale | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in muscle spasticity of the upper extremity
Change from baseline in the Motricity Index (upper extremity) | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in muscle power of the paretic upper extremity.
Change from baseline in cancellation tests (single letter, number, bells) | Baseline, End (4-6 weeks) and 4-weeks follow-up
  Assessment of change from baseline in visual scanning deficits

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Bermudez i Badia, PhD, Principal Investigator — Universidade da Madeira
Locations (1):
- SESARAM, Funchal, Madeira, Portugal

REFERENCES:
- [Background] Cameirao MS, Faria AL, Paulino T, Alves J, Bermudez I Badia S. The impact of positive, negative and neutral stimuli in a virtual reality cognitive-motor rehabilitation task: a pilot study with stroke patients. J Neuroeng Rehabil. 2016 Aug 9;13(1):70. doi: 10.1186/s12984-016-0175-0. PMID 27503215